CLINICAL TRIAL: NCT01927250
Title: Influence of Multi-dimensional Wellness Program (Diet, Art and Biofield Therapy) on Quality of Life in Japanese Population
Brief Title: Influence of Multi-dimensional Wellness Program on Quality of Life
Acronym: MDWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MOA Health Science Foundation (Other)
Responsible Party: Principal Investigator, Kiyoshi Suzuki, President, MOA Health Science Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MOA-003
Record Dates: First submitted 2013-08-17; First posted 2013-08-22 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Healthy; Physical Disorders; Mental Disorders
Keywords: cohort study; diet program; art therapy; laying-on-of-hands; quality of life
MeSH Terms: conditions — Mental Disorders | interventions — Health Promotion; Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Okada Health and Wellness program (Experimental): 12,166 Japanese volunteers with/without illness, who were interested in practicing Okada Health and Wellness program for 3 consecutive months.
  Interventions: Behavioral: Okada Health and Wellness program

INTERVENTIONS:
Behavioral: Okada Health and Wellness program — Each participant were encouraged to practice the diet program and art therapy established by the MOA International Corporation, and to receive Okada Purifying Therapy, a domain of biofield therapy, for 3 consecutive months.
  Other Names: diet program; art therapy; biofield therapy

SUMMARY:
The purpose of this study is to determine whether multi-dimensional wellness program (diet, art and biofield therapy) influences the quality of life for those with different health status in Japan.

DETAILED DESCRIPTION:
Combination of wellness programs may be one of the best approaches to improve quality of life; however, the effectiveness of a treatment that combines various programs is also yet to be clarified. This study investigated the influence of Okada Health and Wellness program on the quality of life for healthy people and those with illness in Japan. Okada Health and Wellness program consists of 3 components: diet, art and biofield therapy.

ELIGIBILITY:
Inclusion Criteria:

* Those who were interested in practicing the diet program and art therapy established by the MOA International Corporation.
* Able to receive Okada Purifying Therapy, a domain of biofield therapy at least once a week.
* Competent to answer the Japanese questionnaires for quality of life
* Aged 16 years or older

Exclusion Criteria:

* Those who did not match the inclusion criteria

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12166 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
change of quality of life | baseline and after 3 months
  Participants were encouraged to practice Okada Health and Wellness program during the intervention period (3 months). They completed a quality of life questionnaire before and after the intervention period.

SECONDARY OUTCOMES:
Adjusted odds ratios of the factors associated with the change of quality of life. | in 1 year
  After collecting all the eligible data, to be clarified are such personal variables as demographic factors and the 3 components of Okada Health and Wellness program that influence the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Suzuki, MD, PhD, Principal Investigator — MOA Health Science Foundation
Locations (1):
- MOA Health Science Foundation, Tokyo, Japan

REFERENCES:
- [Derived] Suzuki K, Kimura T, Uchida S, Katamura H, Tanaka H. The Influence of a Multimodal Health Program with Diet, Art, and Biofield Therapy on the Quality of Life of People in Japan. J Altern Complement Med. 2019 Mar;25(3):336-345. doi: 10.1089/acm.2018.0291. Epub 2019 Feb 11. PMID 30742776
- See also: Click here for more information about activities of MOA Health Science Foundation (Japanese) — http://www.mhs.or.jp
- See also: Click here for more information about Okada Health and Wellness program, a multi-dimensional wellness program — http://www.moainternational.or.jp